CLINICAL TRIAL: NCT01526603
Title: High Dose Chemotherapy and Autologous Peripheral Blood Stem Cell (PBSC) Rescue for Neuroblastoma: Standard of Care Considerations
Brief Title: High Dose Chemotherapy and Autologous Transplant for Neuroblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011OC072; MT2011-11C (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Neuroblastoma
Keywords: peripheral blood stem cell transplantation; autologous stem cell transplant
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Granulocyte Colony-Stimulating Factor; Radiotherapy; Isotretinoin; Melphalan; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Treated for Neuroblastoma (Other): According to patient weight and renal function, consolidation chemotherapy using various doses of Melphalan, Etoposide, and Carboplatin followed by autologous stem cell infusion and serial post-transplant Granulocyte Colony Stimulating Factor, radiation therapy and Isotretinoin maintenance therapy.
  Interventions: Drug: Carboplatin; Biological: Autologous stem cell infusion; Biological: Granulocyte colony stimulating factor; Radiation: Radiation therapy; Drug: Isotretinoin (13-cis-retinoic acid); Drug: Melphalan; Drug: Etoposide

INTERVENTIONS:
Drug: Carboplatin — Carboplatin intravenously (IV), 425 mg/m2/dose (or if ≤ 12kg, 14.2 mg/kg/dose) once daily x 4 doses on days 7 through 4 pretransplant.
  Other Names: Paraplatin
Biological: Autologous stem cell infusion — On day 0 the stem cells will be infused immediately after thawing over 15-60 minutes per institutional guidelines.
Biological: Granulocyte colony stimulating factor — Beginning on day 0 after infusion of the PBSC, patients will receive G-CSF subcutaneously (SQ) or IV (SQ preferred) 5 micrograms/kg once daily and continuing once daily until post-nadir absolute neutrophil count (ANC) > 2000/μL for 3 consecutive days.
  Other Names: G-CSF
Radiation: Radiation therapy — It is suggested that patients who have a complete surgical resection of the primary tumor receive 21.6 Gy external beam radiation therapy (EBRT) to the post-induction chemotherapy, pre-operative primary tumor volume. It is suggested that patients who have an incomplete surgical resection of the primary tumor (residual soft tissue mass measuring >1 cm3) will receive 21.6 Gy EBRT to the postinduction chemotherapy, pre-operative primary tumor volume and an additional boost of 14.4 Gy EBRT to the gross residual tumor (total dose 36 Gy to gross residual tumor volume). Radiation should be given after stem cell transplantation and should start no sooner than 28 days post transplant.
Drug: Isotretinoin (13-cis-retinoic acid) — Post-transplant maintenance therapy with cis-RA daily for 14 days every 28 days repeated for 6 months. This phase of the therapy can be initiated by the BMT team and continued by the referring physician. It is recommended to begin Isotretinoin at day 66 post-transplant and no later than day 100. For patients ≤12 kg, isotretinoin (accutane) should be administered at 5.33 mg/kg/dose divided twice daily. For patients >12 kg isotretinoin (accutane) should be administered at 160 mg/m^2/day divided twice a day. Patients should be considered for monoclonal antibody therapy against GD2, such as ch14.18 if such trials are available.
  Other Names: Accutane
Drug: Melphalan — Melphalan Intravenously (IV), 70 mg/m2/dose (or if ≤ 12 kg, 2.3 mg/kg/dose) once daily x 3 doses on days 7 through 5 pretransplant
  Other Names: Alkeran
Drug: Etoposide — Etoposide intravenously (IV), 338 mg/m2/dose (or if ≤ 12kg, 11.3 mg/kg/dose) once daily x 4 doses on days 7 through 4 pretransplant
  Other Names: Eposin; VP-16

SUMMARY:
This is a standard of care document, outlining the therapy for children with high risk neuroblastoma who are not eligible for Children's Oncology Group (COG) studies.

DETAILED DESCRIPTION:
This therapy involves the use of melphalan, etoposide, and carboplatin (consolidation chemotherapy); autologous stem cell rescue, post-transplant radiation therapy and a maintenance phase with Isotretinoin (Accutane, 13-cis-retinoic acid) therapy. If available, patients should also consider post-transplant therapy with cytokines and monoclonal antibody (ch14.18) on a COG or New Approaches to Neuroblastoma Therapy (NANT) trial.

ELIGIBILITY:
Inclusion Criteria:

* Less than 30 years of age at diagnosis of neuroblastoma
* No evidence of disease progression: defined as increase in tumor size of >25% or new lesions
* Recovery from last induction course of chemotherapy (absolute neutrophil count > 500 and platelet > 20,000)
* No uncontrolled infection
* Minimum frozen peripheral blood stem cells (PBSCs) of 2 x 10^6 CD34 cells/kg for transplant are mandatory and 2 x 10^6 CD34 cells/kg for back-up are strongly recommended (thus, PBSC of 4 x 106 CD34 cells/kg is encouraged)
* Adequate organ function defined as:

  * Hepatic: aspartate aminotransferase (AST) < 3 x upper limit of institutional normal 8 Cardiac: shortening fraction ≥ 27% or ejection fraction ≥ 50%, no clinical congestive heart failure 8 Renal: Creatinine clearance or glomerular filtration rate (GFR) > 60 mL/min/1.73m^2 If a creatinine clearance is performed at end induction and the result is < 100 ml/min/1.73m^2, a GFR must then be performed using a nuclear blood sampling method or iothalamate clearance method. Camera method is NOT allowed as measure of GFR prior to or during Consolidation therapy for patients with GFR or creatinine clearance of < 100 ml/min/1.73m^2

Exclusion Criteria

* Patients with progressive disease should consider participating in phase I studies since consolidation therapy using the regimen outlined in this document have not been determined to be useful.
* Patients who are delayed in consolidation chemotherapy beyond 8 weeks, and don't meet organ function criteria.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Successful Engraftment | Day 42
  The time to neutrophil engraftment will be assessed by standard statistical approaches.

SECONDARY OUTCOMES:
Number of Patients with Disease Free Survival | 2 Years
  The number of patients alive and disease free will be assessed using standard statistical approaches.
Overall Survival | 2 Years
  The number of patients alive will be assessed by standard statistical approaches.
Number of Patients with Treatment Related Death | 1 Year
  The rate of treatment related mortality will be assessed by cumulative incidence approach.
Number of Patients with Disease Free Survival | 5 Years
  The number of patients alive and disease free will be assessed using standard statistical approaches.
Overall Survival | 5 Years
  The number of patients alive will be assessed by standard statistical approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Gupta, MBBS, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States